CLINICAL TRIAL: NCT01380158
Title: Preventing Preterm Birth With a Pessary
Acronym: PrePPy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-225
Record Dates: First submitted 2011-06-15; First posted 2011-06-27 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2011-06

CONDITIONS: Preterm Birth
Keywords: pessary; preterm birth; short cervix; cervical incompetence
MeSH Terms: conditions — Premature Birth; Uterine Cervical Incompetence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pessary use during pregnancy (Experimental): Device: Cup pessary
  Interventions: Device: Cup pessary (Bioteque America, Inc)
- Expectant management (No Intervention): Expectant Management + weekly intramuscular progesterone injections

INTERVENTIONS:
Device: Cup pessary (Bioteque America, Inc) — Placement of cup pessary in the vagina after randomization
  Arms: Pessary use during pregnancy

SUMMARY:
The primary objective of this study, is to determine the effect of a Cup pessary, a device that is currently readily available in the USA and similar in design to the Arabin pessary, on the incidence of delivery prior to 37 weeks in women with a history of prior spontaneous birth (before 37 weeks) and incidentally found to have a cervix less than 25 mm in length prior to 23 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies in patients with a history of spontaneous preterm birth (previous delivery between 17 0/7 weeks and 36 6/7 weeks).
* Women ages 18 to 45 years of age

Exclusion Criteria:

* Major fetal abnormalities (defined as those that are lethal or require prenatal or postnatal surgery), fetal death, or fetal growth restriction diagnosed before randomization.
* Presence of prophylactic cervical cerclage
* Significant maternal-fetal complications (treated chronic hypertension, insulin dependant diabetes mellitus, red cell isoimmunization)
* Painful regular uterine contractions, or ruptured membranes
* Visual cervical dilation of 2cm or greater and visible membranes.
* Patients with a pregnancy dated by an ultrasound after 20 weeks gestation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
delivery prior to 37 weeks of gestation | within the first 30 days after delivery of the neonate
  Gestational age at birth will be recorded

SECONDARY OUTCOMES:
Rate of birth less than seven days from randomization | within the first 30 days after delivery of the neonate
  Gestational age at birth will be recorded
Previable birth (<24 weeks) | within the first 30 days after delivery of the neonate
  Gestational age at birth will be recorded
Perinatal death | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  defined as either a stillbirth or postnatal death prior to hospital discharge
Low birth weight | within the first 30 days after delivery of the neonate
  Birthweight at delivery will be recorded
Major adverse neonatal outcomes | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  intraventricular hemorrhage, respiratory distress syndrome of the newborn, retinopathy of prematurity, or necrotizing enterocolitis
Need for neonatal special care | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  ventilation, phototherapy, treatment for sepsis, blood transfusion
Incidence of complications due to pessary | Every 4 weeks while pregnant with pessary in situ
  Incidence of bacterial vaginosis, urinary tract infections, vaginal erosions will be recorded at monthly visits.

CONTACTS AND LOCATIONS:
Overall Officials: Rita W Driggers, MD, Principal Investigator — Medstar Health Research Institute
Locations (3):
- United States (3):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Franklin Square Hospital, Baltimore, Maryland

REFERENCES:
- [Background] Iams JD, Goldenberg RL, Meis PJ, Mercer BM, Moawad A, Das A, Thom E, McNellis D, Copper RL, Johnson F, Roberts JM. The length of the cervix and the risk of spontaneous premature delivery. National Institute of Child Health and Human Development Maternal Fetal Medicine Unit Network. N Engl J Med. 1996 Feb 29;334(9):567-72. doi: 10.1056/NEJM199602293340904. PMID 8569824
- [Background] Owen J, Hankins G, Iams JD, Berghella V, Sheffield JS, Perez-Delboy A, Egerman RS, Wing DA, Tomlinson M, Silver R, Ramin SM, Guzman ER, Gordon M, How HY, Knudtson EJ, Szychowski JM, Cliver S, Hauth JC. Multicenter randomized trial of cerclage for preterm birth prevention in high-risk women with shortened midtrimester cervical length. Am J Obstet Gynecol. 2009 Oct;201(4):375.e1-8. doi: 10.1016/j.ajog.2009.08.015. PMID 19788970
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] Vitsky M. Pessary treatment of the incompetent cervical os. Obstet Gynecol. 1968 May;31(5):732-3. doi: 10.1097/00006250-196805000-00024. No abstract available. PMID 5646408
- [Background] Oster S, Javert CT. Treatment of the incompetent cervix with the Hodge pessary. Obstet Gynecol. 1966 Aug;28(2):206-8. doi: 10.1097/00003081-196608000-00011. No abstract available. PMID 5944837
- [Background] Arabin B, Halbesma JR, Vork F, Hubener M, van Eyck J. Is treatment with vaginal pessaries an option in patients with a sonographically detected short cervix? J Perinat Med. 2003;31(2):122-33. doi: 10.1515/JPM.2003.017. PMID 12747228
- [Background] Antczak-Judycka A, Sawicki W, Spiewankiewicz B, Cendrowski K, Stelmachow J. [Comparison of cerclage and cerclage pessary in the treatment of pregnant women with incompetent cervix and threatened preterm delivery]. Ginekol Pol. 2003 Oct;74(10):1029-36. Polish. PMID 14669390